CLINICAL TRIAL: NCT02585934
Title: A Phase 3, Double-blind, Randomized Study of RVT-101 Versus Placebo When Added to Existing Stable Donepezil Treatment in Subjects With Mild to Moderate Alzheimer's Disease
Brief Title: Study Evaluating Intepirdine (RVT-101) in Subjects With Mild to Moderate Alzheimer's Disease on Donepezil: MINDSET Study
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Axovant Sciences Ltd. (Industry)
Responsible Party: Sponsor
Organization: Sio Gene Therapies (Industry)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: RVT-101-3001
Record Dates: First submitted 2015-10-22; First posted 2015-10-26 (Estimated); Results first posted 2018-12-05 (Actual); Last update posted 2018-12-05 (Actual); Status verified 2018-11

CONDITIONS: Alzheimer's Disease
Keywords: Alzheimer's disease; RVT-101; donepezil; intepirdine; dementia
MeSH Terms: conditions — Alzheimer Disease; Dementia | interventions — 3-benzenesulfonyl-8-piperazin-1-ylquinoline

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- RVT-101 (Experimental): RVT-101 adjunct to 5 mg or 10 mg donepezil
  Interventions: Drug: RVT-101
- Placebo (Placebo Comparator): Placebo adjunct to 5 mg or 10 mg donepezil
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: RVT-101 — once daily, oral, 35 mg tablets
  Arms: RVT-101
Drug: Placebo — once daily, oral, pill manufactured to match RVT-101 35 mg tablet
  Arms: Placebo

SUMMARY:
This study seeks to confirm a demonstrated treatment effect of intepirdine (RVT-101) as an adjunctive therapy to donepezil for the treatment of subjects with Alzheimer's disease.

DETAILED DESCRIPTION:
This Phase 3 study seeks to confirm a demonstrated treatment effect of intepirdine (RVT-101) on both cognition and activities of daily living when added to stable donepezil treatment in subjects with mild-to-moderate Alzheimer's disease after 24 weeks of double-blind treatment. This study will also provide further information on the safety and tolerability of the 35-mg dose of intepirdine (RVT-101) when used in combination with donepezil compared to donepezil alone. This study is being conducted under the agreement of a Special Protocol Assessment by FDA. Subjects completing this study will be eligible to enroll in a 12 month open-label study of RVT-101 (RVT-101-3002) in which concomitant medications for the treatment of Alzheimer's disease including memantine will be allowed.

ELIGIBILITY:
Inclusion Criteria:

* Male or female subject with AD
* Ongoing donepezil therapy for AD
* An MMSE score 12 to 24 inclusive at Screening; MMSE score 10-26 inclusive at Baseline
* Hachinski Ischaemia score less than or equal to 4 at Screening.
* If female, subject must be: a. of non-childbearing potential or surgically sterile; or, b. willing to use an adequate methods of birth control. Male subjects who are sexually active will also be required to use an adequate form of birth control.
* Subject has the ability to comply with procedures for cognitive and other testing in the opinion of the investigator.
* Subject has a reliable caregiver who is willing to report on subject's status throughout the study.

Exclusion Criteria:

Other Causes for Dementia

* Diagnosis of vascular dementia
* Atypical clinical features or clinical course of dementia that would lead the investigator to conclude symptoms are more likely due to an alternate dementia diagnosis including, but not limited to, frontotemporal dementia, Lewy body dementia, or others.

Confounding Medical Conditions

* History of significant psychiatric illness such as schizophrenia or bipolar affective disorder or any other significant psychiatric illness that in the opinion of the investigator would interfere with participation in the study;
* Any clinically relevant concomitant disease, which, in the opinion of the investigator, makes the subject unsuitable for inclusion in the study.

Ages: 50 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1315 (Actual)
Dates: Start 2015-10 (Actual); Primary Completion 2017-09 (Actual); Study Completion 2017-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ilise Lombardo, MD, Study Director — Axovant Sciences, Inc., Vice President, Clinical Research
Locations (197):
- United States (61):
  - US112, Phoenix, Arizona
  - US220, Tucson, Arizona
  - US168, Encino, California
  - US117, Fullerton, California
  - US214, Los Angeles, California
  - US189, Pasadena, California
  - US096, Rancho Mirage, California
  - US0195, Santa Ana, California
  - US016, Simi Valley, California
  - US106, Temecula, California
  - US179, Hamden, Connecticut
  - US171, Norwich, Connecticut
  - US088, Atlantis, Florida
  - US007, Brooksville, Florida
  - US002, Hallandale, Florida
  - US140, Hialeah, Florida
  - US216, Miami, Florida
  - US110, Miami, Florida
  - US172, North Palm Beach, Florida
  - US003, Orlando, Florida
  - US256, Pensacola, Florida
  - US037, Tampa, Florida
  - US042, Tampa, Florida
  - US004, The Villages, Florida
  - US048, Atlanta, Georgia
  - US046, Atlanta, Georgia
  - US217, Columbus, Georgia
  - US111, Baton Rouge, Louisiana
  - US095, Shreveport, Louisiana
  - US116, Newton, Massachusetts
  - US174, Quincy, Massachusetts
  - US144, Hattiesburg, Mississippi
  - US094, Las Vegas, Nevada
  - US135, Berlin, New Jersey
  - US197, Lawrenceville, New Jersey
  - US215, Mount Arlington, New Jersey
  - US057, Paterson, New Jersey
  - US209, Toms River, New Jersey
  - US036, West Long Branch, New Jersey
  - US001, Albany, New York
  - US049, Brooklyn, New York
  - US097, New Hyde Park, New York
  - US177, New Windsor, New York
  - US142, New York, New York
  - US044, New York, New York
  - US150, Chapel Hill, North Carolina
  - US185, Charlotte, North Carolina
  - US113, Beachwood, Ohio
  - US136, Cincinnati, Ohio
  - US008, Cincinnati, Ohio
  - US119, Shaker Heights, Ohio
  - US134, Portland, Oregon
  - US169, Media, Pennsylvania
  - US187, Philadelphia, Pennsylvania
  - US162, Plains, Pennsylvania
  - US148, Willow Grove, Pennsylvania
  - US115, Houston, Texas
  - US043, San Antonio, Texas
  - US143, Orem, Utah
  - US149, Charlottesville, Virginia
  - US170, Spokane, Washington
- Argentina (17):
  - AR130, La Plata, Buenos Aires
  - AR041, La Plata, Buenos Aires
  - AR101, Buenos Aires
  - AR060, Buenos Aires
  - AR084, Ciudad Autónoma de Buenos Aire
  - AR027, Ciudad Autónoma de Buenos Aire
  - AR012, Ciudad Autónoma de Buenos Aire
  - AR160, Ciudad Autónoma de Buenos Aire
  - AR040, Ciudad Autónoma de Buenos Aire
  - AR028, Ciudad Autónoma de Buenos Aire
  - AR081, Ciudad Autónoma de Buenos Aire
  - AR035, Ciudad Autónoma de Buenos Aire
  - AR051, Córdoba
  - AR137, Córdoba
  - AR210, Mendoza
  - AR219, Mendoza
  - AR059, Santiago del Estero
- Australia (6):
  - AU227, Caulfield
  - AU079, Chermside
  - AU032, Heidelberg West
  - AU062, Herston
  - AU011, Hornsby
  - AU138, West Perth
- Bulgaria (4):
  - BU125, Rousse
  - BU131, Sofia
  - BU198, Sofia
  - BU073, Varna
- Canada (10):
  - CA151, Medicine Hat, Alberta
  - CA120, Kamloops, British Columbia
  - CA054, Kelowna, British Columbia
  - CA188, Kelowna, British Columbia
  - CA186, Penticton, British Columbia
  - CA141, West Vancouver, British Columbia
  - CA147, Newmarket, Ontario
  - CA196, North York, Ontario
  - CA237, Toronto, Ontario
  - CA236, Gatineau, Quebec
- Chile (4):
  - CH212, Antofagasta, Antofagasta
  - CH061, Santiago, Santiago Metropolitan
  - CH075, Santiago, Santiago Metropolitan
  - CH076, Santiago, Santiago Metropolitan
- Croatia (5):
  - CR069, Zagreb
  - CR122, Zagreb
  - CR068, Zagreb
  - CR070, Zagreb
  - CR083, Zagreb
- Czechia (5):
  - CZ128, Prague
  - CZ207, Prague
  - CZ132, Prague
  - CZ129, Prague
  - CZ161, Rychnov nad Kněžnou
- France (4):
  - FR231, Lille
  - FR182, Marseille
  - FR221, Paris
  - FR202, Villeurbanne
- Germany (12):
  - GE206, Bad Homburg
  - GE091, Berlin
  - GE071, Berlin
  - GE139, Berlin
  - GE230, Cologne
  - GE252, Ellwangen
  - GE180, Leipzig
  - GE228, Mannheim
  - GE017, München
  - GE157, Nuremberg
  - GE098, Ulm
  - GE251, Westerstede
- Italy (9):
  - IT053, Brescia
  - IT124, Cefalù
  - IT030, Pavia
  - IT103, Perugia
  - IT072, Roma
  - IT183, Roma
  - IT029, Roma
  - IT175, Rome
  - IT085, Torino
- Poland (10):
  - PO013, Bialystok
  - PO024, Bydgoszcz
  - PO010, Bydgoszcz
  - PO107, Katowice
  - PO092, Katowice
  - PO023, Krakow
  - PO025, Krakow
  - PO009, Poznan
  - PO014, Szczecin
  - PO074, Warsaw
- Serbia (7):
  - SE164, Belgrade
  - SE090, Belgrade
  - SE166, Belgrade
  - SE193, Belgrade
  - SE155, Kragujevac
  - SE031, Novi Kneževac
  - SE165, Vršac
- Singapore (2):
  - SI052, Singapore
  - SI026, Singapore
- Slovakia (6):
  - SL056, Banská Bystrica
  - SL192, Bratislava
  - SL200, Dubnica nad Váhom
  - SL191, Košice
  - SL078, Krompachy
  - SL077, Svidník
- South Korea (3):
  - SK066, Busan
  - SK067, Seoul
  - SK190, Seoul
- Spain (12):
  - SP249, Alicante
  - SP176, Barcelona
  - SP022, Barcelona
  - SP021, Barcelona
  - SP250, Barcelona
  - SP019, Ceuta
  - SP194, Donostia / San Sebastian
  - SP222, Getxo
  - SP018, Madrid
  - SP093, Madrid
  - SP184, Sant Cugat del Vallès
  - SP020, Terrassa
- Taiwan (3):
  - TA065, Kaohsiung City
  - TA086, Taipei
  - TA121, Taoyuan District
- United Kingdom (17):
  - UK063, Bath
  - UK038, Blackpool
  - UK233, Cambridge
  - UK033, Cannock
  - UK211, Epping
  - UK234, Guildford
  - UK055, Leeds
  - UK039, London
  - UK034, Manchester
  - UK229, Norwich
  - UK087, Oxford
  - UK235, Plymouth
  - UK100, Sheffield
  - UK064, Southampton
  - UK152, Southampton
  - UK153, Swindon
  - UK154, Warrington

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 2173 participants signed consent and were screened for participation. Of these, 1470 entered a 3-week single-blind placebo run-in period with treatment with placebo qd + stable dose of donepezil 5 or 10 mg qd. There was an overlap between the participants from the run-in period and the participants that were randomized during the treatment period.
Groups:
- RVT-101: RVT-101 adjunct to 5 mg or 10 mg donepezil
  RVT-101: once daily, oral, 35 mg tablets for up to 27 weeks
- Placebo: Placebo adjunct to 5 mg or 10 mg donepezil
  Placebo: once daily, oral, pill manufactured to match RVT-101 35 mg tablet for up to 27 weeks
Period: Overall Study
Arm/Group | RVT-101 | Placebo
Started | 661 | 654
Safety Population (The Safety population included subjects who took at least 1 dose of double-blind study drug) | 656 | 651
Intent to Treat (ITT) (Subjects took at least 1 dose of double-blind study drug and had at least 1 post-baseline assessment) | 643 | 633
Per Protocol (PP) (Subjects in the ITT population who had no major protocol violations) | 603 | 582
Completed (Subjects in the ITT population who completed the study) | 592 | 581
Not Completed | 69 | 73
Not completed — Lost to Follow-up | 2 | 2
Not completed — Protocol Violation | 14 | 11
Not completed — Adverse Event | 21 | 22
Not completed — Physician Decision | 3 | 2
Not completed — Withdrawal by Subject | 7 | 21
Not completed — Lack of Efficacy | 2 | 1
Not completed — Death | 2 | 0
Not completed — Caregiver Withdrew Consent | 7 | 7
Not completed — Sponsor Termination | 1 | 2
Not completed — Another Reason | 10 | 5

BASELINE CHARACTERISTICS:
Population: ITT population
Groups:
- Total: Total of all reporting groups
Arm/Group | RVT-101 | Placebo | Total
Number analyzed (Participants) | 643 | 633 | 1276
Age, Continuous [Mean (Full Range); unit: years] | 72.7 [50 to 85] | 72.5 [50 to 86] | 72.6 [50 to 86]
Age, Customized [Count of Participants; unit: Participants]
  < 74 years | 309 | 312 | 621
  >/= 74 years | 334 | 321 | 655
  < 65 years | 98 | 97 | 195
  >/=65 years | 545 | 536 | 1081
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 386 | 394 | 780
  Male | 257 | 239 | 496
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 120 | 108 | 228
  Not Hispanic or Latino | 518 | 519 | 1037
  Unknown or Not Reported | 5 | 6 | 11
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race: White | 595 | 592 | 1187
  Race: Black or African American | 12 | 10 | 22
  Race: Asian | 27 | 20 | 47
  Race: American Indian or Alaska Native | 0 | 0 | 0
  Race: Native Hawaiian or Other Pacific Islander | 0 | 1 | 1
  Race: Others | 2 | 1 | 3
  Race: Not Applicable | 3 | 5 | 8
  Race: Missing | 4 | 4 | 8
BMI [Mean (Full Range); unit: kg/m^2] — Population: Data was missing for one subject
  kg/m^2
    number analyzed (Participants) | 642 | 633 | 1275
    (all) | 26.4 [17.2 to 56.3] | 26.5 [15.2 to 45.3] | 26.4 [15.2 to 56.3]

OUTCOME MEASURES:

1. Primary Outcome: Alzheimer's Disease Assessment Scale - Cognitive Subscale 11 Items (ADAS-Cog-11) Score Change From Baseline to Week 24
Description: The 11-item ADAS-Cog assesses a range of cognitive abilities including memory, comprehension, orientation in time and place, and spontaneous speech. The ADAS-Cog-11 total score range is from 0 to 70, with a higher score indicating more severe cognitive impairment.
Time Frame: Baseline, 24 weeks
Population: ITT Population with data at both timepoints.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | RVT-101 | Placebo
Number analyzed (Participants) | 584 | 577
units on a scale | 0.39 (0.211) | 0.75 (0.213)
Statistical Analysis 1: Comparison: RVT-101 vs Placebo; Test type: Superiority; p = 0.2249, Mixed Models Analysis — the threshold for statistical significance was p=0.05; Statistical Method: Mixed model for repeated measures; least square mean difference = -0.36, 95% CI 2-sided [-0.95 to 0.22]

2. Primary Outcome: Alzheimer's Disease Cooperative Study - Activities of Daily Living (ADCS-ADL) Score Change From Baseline to Week 24
Description: The ADCS-ADL scale measures functional impairment in terms of activities of daily living. The score ranges from 0 to 78. The lower the score, the greater the impairment; higher scores indicate better (more desirable) function
Time Frame: Baseline, 24 weeks
Population: ITT Population with data at both endpoints
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | RVT-101 | Placebo
Number analyzed (Participants) | 588 | 575
units on a scale | -1.06 (0.289) | -0.97 (0.293)
Statistical Analysis 1: Comparison: RVT-101 vs Placebo; Test type: Superiority; p = 0.8260, Mixed Models Analysis — the threshold for statistical significance was p=0.05; Statistical Method: Mixed model for repeated measures; least square mean difference = -0.09, 95% CI 2-sided [-0.90 to 0.72]

3. Secondary Outcome: Clinical Global Impression of Change - Plus Caregiver Interview (CIBIC+) Score at Week 24
Description: The CIBIC+ assessment measures the global functioning of the subject. The CIBIC+ is scored as a seven-point categorical rating, ranging from a score of 1 (indicating "very much improved"), to a score of 4 (indicating "no change"), or to a score of 7 (indicating "very much worse.") Lower CIBIC+ scores indicate better (more desirable) function
Time Frame: 24 weeks
Population: ITT population at the Week 24 timepoint
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | RVT-101 | Placebo
Number analyzed (Participants) | 577 | 568
units on a scale | 4.18 (0.037) | 4.30 (0.037)
Statistical Analysis 1: Comparison: RVT-101 vs Placebo; Test type: Superiority; p = 0.0234, Mixed Models Analysis — the threshold for statistical significance was p=0.05; Statistical Method: Mixed model for repeated measures; least square mean difference = -0.12, 95% CI 2-sided [-0.22 to -0.02]

4. Secondary Outcome: The Dependence Scale (DS) Score Change From Baseline to Week 24
Description: The DS measures the amount of assistance patients with dementia require in performing daily activities. The scale consists of 13 items, representing a range of severity from mild to severe levels of dependency. The score range is from 0 to 15 with higher scores indicating greater dependency.
Time Frame: Baseline, 24 weeks
Population: ITT population at both timepoints
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | RVT-101 | Placebo
Number analyzed (Participants) | 580 | 568
units on a scale | 0.30 (0.070) | 0.17 (0.071)
Statistical Analysis 1: Comparison: RVT-101 vs Placebo; Test type: Superiority; p = 0.2096, Mixed Models Analysis — the threshold for statistical significance was p=0.05; Statistical Method: Mixed model for repeated measures; least square mean difference = 0.12, 95% CI 2-sided [-0.07 to 0.32]

5. Secondary Outcome: Neuropsychiatric Inventory (NPI) Score Change From Baseline to Week 24
Description: The NPI is a behavior rating scale composed of a 12-item structured interview of the caregiver that is scored from 0 to 144 (the higher the score, the greater the psychiatric disturbance). It assesses 12 behavioral disturbances occurring in dementia patients: delusions, hallucinations, agitation, dysphoria, anxiety, apathy, irritability, euphoria, disinhibition, aberrant motor activity, night-time behavior disturbances, and eating disturbances. Both the frequency and the severity of each behavior are determined.
Time Frame: Baseline and Week 24
Population: ITT Population at both timepoints
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | RVT-101 | Placebo
Number analyzed (Participants) | 583 | 570
units on a scale | -0.08 (0.339) | 0.06 (0.344)
Statistical Analysis 1: Comparison: RVT-101 vs Placebo; Test type: Superiority; p = 0.7650, Mixed Models Analysis — the threshold for statistical significance was p=0.05; Statistical Method: Mixed model for repeated measures; least square mean difference = -0.14, 95% CI 2-sided [-1.09 to 0.80]

6. Secondary Outcome: ADAS-Cog-13 Score Change From Baseline to Week 24
Description: 13-item ADAS-Cog assesses a range of cognitive abilities including memory, comprehension, orientation in time and place, and spontaneous speech. Most items are evaluated by tests, but some are dependent on clinician ratings on a 5-point scale. The ADAS-Cog-13 is the ADAS-Cog-11 with 2 additional items: delayed word recall and total digit cancellation. Scores for the ADAS-Cog-13 range from 0 to 85 with higher scores indicating greater dysfunction.
Time Frame: Baseline, 24 weeks
Population: ITT at both timepoints
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | RVT-101 | Placebo
Number analyzed (Participants) | 583 | 576
units on a scale | 0.26 (0.233) | 0.64 (0.236)
Statistical Analysis 1: Comparison: RVT-101 vs Placebo; Test type: Superiority; p = 0.2472, Mixed Models Analysis — the threshold for statistical significance was p=0.05; Statistical Method: Mixed model for repeated measures; least square mean difference = -0.38, 95% CI 2-sided [-1.03 to 0.27]

7. Secondary Outcome: Measurement of Concentrations of RVT-101 (Intepirdine) in Plasma
Description: Measurement collected at timepoints Week 6, Week 12, Week 18, and Week 24
Time Frame: Week 6, Week 12, Week 18, Week 24
Population: PK population at specified timepoints: Week 6, Week 12, Week 18, and Week 24
Measure: Geometric Mean (95% Confidence Interval); unit: ng/mL
Arm/Group | RVT-101
Number analyzed (Participants) | 656
ng/mL
  Summary Statistics at Week 6: number analyzed (Participants) | 563
  Summary Statistics at Week 6 | 201.11 [191.88 to 210.78]
  Summary Statistics at Week 12: number analyzed (Participants) | 579
  Summary Statistics at Week 12 | 170.95 [164.40 to 177.76]
  Summary Statistics at Week 18: number analyzed (Participants) | 454
  Summary Statistics at Week 18 | 198.69 [189.36 to 208.48]
  Summary Statistics at Week 24: number analyzed (Participants) | 562
  Summary Statistics at Week 24 | 193.36 [184.60 to 202.53]

ADVERSE EVENTS:
Time Frame: Screening through post treatment (up to 33 weeks)
Groups:
- RVT-101 Treatment: RVT-101 adjunct to 5 mg or 10 mg donepezil
  RVT-101: once daily, oral, 35 mg tablets for up to 27 weeks
- Placebo Treatment: Placebo adjunct to 5 mg or 10 mg donepezil
  Placebo: once daily, oral, pill manufactured to match RVT-101 35 mg tablet for up to 27 weeks
- Screening Period: Participants screened (0-4 weeks) prior to entering to the first dose of single-blind study medication (ie, prior to the Run-In period)
- Run-In Period: Placebo adjunct to 5 mg or 10 mg donepezil
  Placebo: once daily, oral, pill manufactured to match RVT-101 35 mg tablet (for 3 weeks)
- RVT-101 Post-Treatment; Placebo Post-Treatment: Subjects reported adverse events after completing the treatment period.
  The Post-Treatment period - defined as up to 30 days post-last-dose
Arm/Group | RVT-101 Treatment | Placebo Treatment | Screening Period | Run-In Period | RVT-101 Post-Treatment | Placebo Post-Treatment
All-Cause Mortality (participants affected / at risk) | 3/656 | 2/651 | 1/2173 | 1/1470 | 0/656 | 1/651
Serious Adverse Events (participants affected / at risk) | 40/656 | 44/651 | 12/2173 | 14/1470 | 3/656 | 3/651
Other Adverse Events (participants affected / at risk) | 191/656 | 166/651 | 0/2173 | 0/1470 | 0/656 | 0/651
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | RVT-101 Treatment (N=656) | Placebo Treatment (N=651) | Screening Period (N=2173) | Run-In Period (N=1470) | RVT-101 Post-Treatment (N=656) | Placebo Post-Treatment (N=651)
Cerebrovascular Accident (Nervous system disorders) | 0 | 3 | 0 | 0 | 0 | 0
Syncope (Nervous system disorders) | 2 | 1 | 0 | 0 | 0 | 0
Transient ischaemic attack (Nervous system disorders) | 2 | 1 | 1 | 0 | 1 | 0
Ischaemic stroke (Nervous system disorders) | 2 | 0 | 0 | 0 | 0 | 0
Seizure (Nervous system disorders) | 0 | 2 | 0 | 0 | 0 | 0
Dementia (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0
Dizziness (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0
Headache (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0
Hypoxic-ischaemic encephalopathy (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0
Lethargy (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0
Status epilepticus (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 3 | 0 | 3 | 0 | 0
Acoustic neuroma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0 | 0 | 0
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0 | 0 | 0
Hepatocellular carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0 | 0 | 0
Lung neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0 | 0 | 0
Malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 1 | 0 | 0 | 0
Meningioma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0 | 0 | 0
Ovarian cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0 | 0 | 0
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0 | 0 | 0
Squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 1 | 0 | 0
Uterine leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0 | 0 | 0
Myocardial infarction (Cardiac disorders) | 1 | 2 | 0 | 0 | 0 | 0
Atrial Fibrillation (Cardiac disorders) | 1 | 1 | 0 | 0 | 0 | 0
Angina pectoris (Cardiac disorders) | 0 | 1 | 0 | 0 | 0 | 0
Angina unstable (Cardiac disorders) | 0 | 1 | 0 | 0 | 0 | 0
Atrioventricular block (Cardiac disorders) | 0 | 1 | 1 | 0 | 0 | 0
Cardiac arrest (Cardiac disorders) | 0 | 1 | 0 | 0 | 0 | 0
Cardiac failure congestive (Cardiac disorders) | 0 | 1 | 0 | 0 | 0 | 0
Cardio-respiratory arrest (Cardiac disorders) | 1 | 0 | 0 | 0 | 0 | 0
Mitral valve prolapse (Cardiac disorders) | 0 | 1 | 0 | 0 | 0 | 0
Pericardial effusion (Cardiac disorders) | 1 | 0 | 0 | 0 | 0 | 0
Right ventricular failure (Cardiac disorders) | 1 | 0 | 0 | 0 | 0 | 0
Sinus node dysfunction (Cardiac disorders) | 1 | 0 | 0 | 1 | 0 | 0
Diverticulitis (Infections and infestations) | 2 | 2 | 0 | 1 | 0 | 0
Pneumonia (Infections and infestations) | 2 | 1 | 0 | 0 | 0 | 0
Urinary tract infection (Infections and infestations) | 1 | 1 | 1 | 0 | 0 | 0
Appendicitis (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0
Cellulitis (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0
Gastroenteritis (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0
Fall (Injury, poisoning and procedural complications) | 1 | 3 | 1 | 1 | 0 | 0
Hip fracture (Injury, poisoning and procedural complications) | 1 | 3 | 2 | 0 | 0 | 0
Contusion (Injury, poisoning and procedural complications) | 0 | 1 | 1 | 0 | 0 | 0
Patella fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0 | 0
Pelvic fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0 | 0
Stoma obstruction (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0 | 0
Subdural haematoma (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0 | 0
Upper limb fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0 | 0
Wrist fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0 | 0
Duodenal vascular ectasia (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0
Pancreatitis acute (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0
Proctitis (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0
Small intestinal obstruction (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0
Aggression (Psychiatric disorders) | 1 | 0 | 0 | 0 | 0 | 0
Delirium (Psychiatric disorders) | 1 | 0 | 0 | 0 | 0 | 0
Mental status changes (Psychiatric disorders) | 0 | 1 | 0 | 0 | 0 | 0
Mood altered (Psychiatric disorders) | 0 | 1 | 0 | 0 | 0 | 0
Psychotic disorder (Psychiatric disorders) | 0 | 1 | 0 | 1 | 0 | 0
Somatic symptom disorder (Psychiatric disorders) | 1 | 0 | 0 | 0 | 0 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 0 | 0 | 0 | 0
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 0
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1 | 1 | 0 | 1
Chest pain (General disorders) | 1 | 0 | 0 | 0 | 0 | 0
Hypothermia (General disorders) | 0 | 1 | 0 | 0 | 0 | 0
Non-cardiac chest pain (General disorders) | 0 | 1 | 0 | 0 | 0 | 0
Inner ear disorder (Ear and labyrinth disorders) | 0 | 1 | 0 | 0 | 0 | 0
Vertigo positonal (Ear and labyrinth disorders) | 1 | 0 | 0 | 0 | 0 | 0
Bile duct stone (Hepatobiliary disorders) | 1 | 0 | 0 | 0 | 0 | 0
Cholecystitis (Hepatobiliary disorders) | 0 | 1 | 0 | 0 | 0 | 0
Hypertension (Vascular disorders) | 0 | 1 | 0 | 0 | 0 | 0
Poor peripheral circulation (Vascular disorders) | 1 | 0 | 0 | 0 | 0 | 0
Haemoglobin decreased (Investigations) | 1 | 0 | 0 | 0 | 0 | 0
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0
Acute kidney injury (Renal and urinary disorders) | 1 | 0 | 0 | 0 | 0 | 0
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 1 | 0 | 0 | 0 | 0 | 0
Humerus fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0 | 0
Cardiac failure (Cardiac disorders) | 0 | 0 | 1 | 0 | 0 | 0
Anaemia (Blood and lymphatic system disorders) | 0 | 0 | 1 | 0 | 0 | 0
Volvulus (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0
lower respiratory tract infection (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0
Squamous cell carcinoma of skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1 | 0 | 0
Infected bite (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0
Foot fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0 | 0
Pubis fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0 | 0
Agitation (Psychiatric disorders) | 0 | 0 | 0 | 1 | 0 | 0
Pneumothorax spontaneous (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 0
Asthenia (General disorders) | 0 | 0 | 0 | 1 | 0 | 0
Dehydration (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 0 | 0
Hydrocephalus (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0
Gait disturbance (General disorders) | 0 | 0 | 0 | 0 | 1 | 0
Sepsis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1
invasive ductal breast carcinoma (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | RVT-101 Treatment (N=656) | Placebo Treatment (N=651) | Screening Period (N=2173) | Run-In Period (N=1470) | RVT-101 Post-Treatment (N=656) | Placebo Post-Treatment (N=651)
Fall (Injury, poisoning and procedural complications) | 37 | 29 | 0 | 0 | 0 | 0
Urinary tract infection (Infections and infestations) | 25 | 26 | 0 | 0 | 0 | 0
Nasopharyngitis (Respiratory, thoracic and mediastinal disorders) | 23 | 19 | 0 | 0 | 0 | 0
Headache (Nervous system disorders) | 17 | 18 | 0 | 0 | 0 | 0
Dizziness (Nervous system disorders) | 19 | 12 | 0 | 0 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 13 | 17 | 0 | 0 | 0 | 0
Nausea (Gastrointestinal disorders) | 17 | 13 | 0 | 0 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 11 | 15 | 0 | 0 | 0 | 0
Bronchitis (Respiratory, thoracic and mediastinal disorders) | 14 | 10 | 0 | 0 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 15 | 7 | 0 | 0 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
All proposed manuscripts, publications or abstracts must be reviewed and approved by the Sponsor 60 days prior to submission for publication. All confidential information identified by the Sponsor must be deleted prior to submission.

DOCUMENTS (3):
  • Study Protocol: Protocol (2016-04-13): https://cdn.clinicaltrials.gov/large-docs/34/NCT02585934/Prot_000.pdf
  • Statistical Analysis Plan: Statistical Analysis Plan Document (2017-08-09): https://cdn.clinicaltrials.gov/large-docs/34/NCT02585934/SAP_001.pdf
  • Statistical Analysis Plan: Statistical Analysis Plan Addendum Document (2017-09-19): https://cdn.clinicaltrials.gov/large-docs/34/NCT02585934/SAP_002.pdf